CLINICAL TRIAL: NCT00347659
Title: Phase 1 Study of the Biologic Lung Volume Reduction (BLVR) System in Patients With Advanced Upper Lobe Predominant Emphysema
Brief Title: US 10 mL Biologic Lung Volume Reduction (BLVR) Phase 1 Emphysema Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Edward Ingenito, MD, PhD, Medical Director &CSO, Aeris Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-C06-001
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Pulmonary Emphysema
Keywords: Lung volume reduction; Bronchoscopy; Emphysema; COPD; NETT; Lung disease; COLD; BLVR
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Treatment (Experimental): Experimental Treatment
  Interventions: Drug: BLVR System

INTERVENTIONS:
Drug: BLVR System — Treatment is administered in a single treatment session.

SUMMARY:
The purpose of this study is to evaluate the safety of the Biologic Lung Volume Reduction System (BLVR) for patients with advanced emphysema.

DETAILED DESCRIPTION:
Emphysema is a progressive, debilitating disease that affects nearly 3 million people in the United States or roughly one percent of the US population. The disease is characterized by destruction of lung tissue as a result of inflammation caused by exposure to noxious inhaled agents for extended periods. The most common cause of this condition is cigarette smoking, although genetic and occupational causes account for up to 10% of cases. Despite aggressive public health initiatives aimed at discouraging the use of cigarettes, smoking-related lung diseases remain a significant cause of disability and death in the United States. Currently there are 46 million smokers in the US. Due to the number of current and new smokers, emphysema is expected to remain a leading cause of morbidity and mortality in the United States for years to come.

Aeris has developed a novel bronchoscopic system for achieving the benefits of lung volume reduction without surgery. The Biologic Lung Volume Reduction (BLVR) System, a new investigational therapy for emphysema, is intended to reduce lung volume over a period of weeks by collapsing and promoting the remodeling of diseased areas of the lung. The resulting reduction in lung volume is intended to restore a more normal physiological relationship between lung and chest wall, improve breathing and exercise capacity and alleviate symptoms of chronic dyspnea. This study will evaluate the safety of the BLVR System in patients with advanced emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced heterogeneous emphysema
* Age >/= 40
* Clinically significant dyspnea
* Failure of standard medical therapy to relieve symptoms
* Pulmonary function tests with protocol-specified ranges

Exclusion Criteria:

* Alpha-1 protease inhibitor deficiency
* Tobacco use within 16 weeks of initial clinic visit
* Body mass index < 15 kg/m2 or > 35 kg/m@
* Clinically significant asthma, chronic bronchitis or bronchiectasis
* Allergy or sensitivity to tetracycline
* Prior lung volume reduction surgery, prior lobectomy or pneumonectomy, prior lung transplantation, prior endobronchial valve placement, prior airway stent placement or prior pleurodesis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
SAEs - Safety of the procedure from initiation of treatment through hospital discharge. | 1 week post treatment
SAEs - Safety of the treatment through Week 12. | 12 weeks post procedure

SECONDARY OUTCOMES:
SAEs - Safety of the treatment through Week 48. | 48 weeks post treatment
Evaluation of radiologic changes. | 12 weeks post treatment
Improvement in exercise capacity. | 12 weeks post treatment
Improvement in quality of life. | 12 weeks post treatment
Decrease in trapped gas. | 12 weeks post treatment
Improvement in lung function. | 12 weeks post trreatment
Improvement in symptoms. | 12 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Temple University Lung Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835